CLINICAL TRIAL: NCT03154931
Title: Group Compassion Focused Therapy for Posttraumatic Stress Disorder
Brief Title: Efficacy of Compassion Focused Therapy in Group for Posttraumatic Stress Disorder
Acronym: GCFT-PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Francisco Lotufo Neto, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Group CFT treatment for PTSD
Record Dates: First submitted 2015-09-24; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: PTSD
Keywords: PTSD; CBT; CFT; compassion; shame; guilty; self-criticism
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-SG (Active Comparator): This CBT-Supportive group will focus on the interaction here-and-now, realizing that the group acts as a secure place, driven by interactions among its participants and therapist and co-therapist. The main objective is to welcome and support the participation of all patients and stimulate the group's initiatives, encouraging interpersonal interactions and mutual aid. There will be no specific therapeutic intervention in relation to any PTSD related content.
  Interventions: Other: CBT-SG
- CFT-G (Experimental): This CFT-group will focus on activities using specific therapeutic strategies, to learn and training compassionate skills - psychoeducation and exercises developed for use in session and at home.They will learn What is compassion and shame? Steps to the training of compassion and how Building a compassionate image. Will use Thoughts Daily Record - self critical and self compassionate. Explanation of Formulation of Strategy Threats and Security, The Three Emotional regulation systems and PTSD formulation - based on shame and guilt. They will learn how to incorporate these skills to everyday situations. At the end, will write an Autobiography writing about this experience and share with the group.
  Interventions: Other: CFT-G

INTERVENTIONS:
Other: CBT-SG — To support the group.
  Arms: CBT-SG
Other: CFT-G — Teach compassionate skills.
  Arms: CFT-G

SUMMARY:
The purpose of this study is to determine the efficacy of a 8-week program of Compassion Focused Therapy in Group comparing to Supportive Cognitive Behavioral Therapy in Group for patients with Posttraumatic Stress Disorder.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial with two parallel groups, with two models of treatment: Group 1 - Control Group - will receive CBT Supportive Group (CBT-SG) and Group 2 - Experimental Group - will receive Compassion Focused Therapy (CFT-G). Will be attended in total, the maximum of 80 patients, with 40 patients in each arm (CBT-SG versus CFT-G). Both groups will be formed by at least eight patients and a maximum of twelve patients who receive eight weekly sessions with an hour and a half each session, and the total duration of treatment will be eight weeks. The groups will be closed, that is, after the start will not be permitted to input any more participants. The experimental group (CFT-G) will be structured and the control group (CBT-SG) will be unstructured, and free format.

All patients will be assessed through self-report scales, within three distinct phases: Assessment I - Initial (before therapy); Assessment II - Final (after therapy); Assessment III - Follow-up (after 3 months of therapy ending).

All groups will be led by a principal therapist and co-therapist. All sessions will be recorded for later evaluation of the researcher responsible for the research.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Administered PTSD Scale 5 Monthly version Criteria A and >30 points

Exclusion Criteria:

* Suicidal patients and/or severe automutilation behavior and/or psychotic symptoms and/or lack of event memory.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Administered Posttraumatic Stress 5 | up to 8 weeks
  40% decrease

SECONDARY OUTCOMES:
Davidson Trauma Scale | up to 8 weeks
  40% decrease
Beck Depression Inventory | up to 8 weeks
  final rating <20.
Beck Anxiety Inventory | up to 8 weeks
  final rating <19.
Beck Hopelessness Scale | up to 8 weeks
  final rating <9.
Self Compassion Scale | up to 8 weeks
  50% increase
Other as a Shame Scale | up to 8 weeks
  50% decrease
Functions of Self Critical Scale | up to 8 weeks
  50% decrease
Connor Davidson Resilience | up to 8 weeks
  50% increase
Outcome Questionnaire 45 | up to 8 weeks
  50% decrease

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Lotufo Neto, PhD, Study Director — University of Sao Paulo General Hospital
Locations (1):
- AMBAN - Anxiety Program at IPQ-HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided